CLINICAL TRIAL: NCT02257294
Title: A Randomised, Double Blind, Placebo-controlled, Parallel Group Trial of Low-dose Adjunctive alTeplase During prIMary PCI
Brief Title: A Trial of Low-dose Adjunctive alTeplase During prIMary PCI
Acronym: T-TIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GN12CA450; 12/170/45 (Other Grant/Funding Number: EME)
Record Dates: First submitted 2014-09-26; First posted 2014-10-06 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Arm (Placebo Comparator): two placebo vials
  Interventions: Other: Placebo
- Arm A (Active Comparator): Alteplase 10mg and placebo vial
  Interventions: Drug: Alteplase; Other: Placebo
- Arm B (Active Comparator): Alteplase 10mg and alteplase 10mg
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Single treatment consisting of a single slow infusion administration after reperfusion with aspiration thrombectomy ± angioplasty but before stenting during primary PCI.
  Other Names: Actilyse
  Arms: Arm A; Arm B
Other: Placebo — Single treatment consisting of a single slow infusion administration after reperfusion with aspiration thrombectomy ± angioplasty but before stenting during primary PCI.
  Arms: Arm A; Control Arm

SUMMARY:
The purpose of this study is to determine the safety and efficacy of reduced doses (10 mg and 20 mg) of intra-coronary alteplase compared with placebo as an adjunct to PCI in reducing MVO and its consequences in high risk patients with STEMI.

DETAILED DESCRIPTION:
Despite numerous interventions, there remains a need to develop new ways to prevent microvascular obstruction (MVO). The investigators aim to select patients with persistent S-T-elevation on the ECG and an occluded artery and heavy thrombus burden at initial angiography. These characteristics are causally linked to MVO. Patients with a thrombotic culprit coronary artery have reduced myocardial perfusion compared to those without and the presence of coronary thrombus is an independent predictor of adverse ischaemic outcomes post-MI. Intra-luminal thrombus, as revealed by intra vascular imaging with optical coherence tomography (OCT) in STEMI patients, has shown that thrombus commonly persists in the culprit coronary artery, including within the stent post-implantation, even when the thrombus is invisible with conventional angiography. The amount of persistent thrombus predicted the likelihood of persistent S-T-segment elevation, a marker of microvascular injury, and impaired perfusion.Therefore, coronary thrombus represents a therapeutic target in primary PCI. The pathophysiology of MVO and microvascular thrombosis has elucidated in MRI studies of reperfused MI in swine. The investigators demonstrated that LATE MVO corresponds closely with infarct zone haemorrhage as revealed by T2-weighted MRI and pathology. The investigators observations were validated by Robbers et al who showed that in swine 7 days post-MI, when LATE MVO and haemorrhage correspond (which is usually the case), there is severe capillary loss and disruption coupled with thrombosis and inflammation. They concluded that following reperfusion, acute inflammation and microvessel thrombosis result in degradation of endothelial integrity and capillary breakdown. Very interestingly, their histology also demonstrated diffuse microvascular thrombosis within the area of late gadolinium enhancement surrounding the haemorrhagic core which explains reduced perfusion (or wash during first pass of gadolinium contrast MRI) within the ischaemic area-at-risk. This observation points to the therapeutic potential of local thrombolysis within the culprit artery circulation.The study addresses the question of whether a pharmacological strategy involving reduced dose alteplase given early during the primary PCI procedure will both prevent and treat distal microvascular thrombosis and MVO and, subsequently, reduce infarct size.Current evidence around the potential safety and efficacy of reduced dose fibrinolysis in primary PCI is limited. These limitations set-the-scene and support the rationale for the clinical trial: Full systemic dose intravenous fibrinolysis to facilitate primary PCI is potentially harmful and increases the risk of off-target bleeding complications; therefore, the investigators will use reduced-dose fibrinolysis. They will directly infuse alteplase into the culprit artery to achieve effective and sustained local plasma concentrations and much lower systemic concentrations of unbound drug. It is anticipated that bleeding rates may be low; therefore, the investigators will measure fibrinogen in all patients. Fibrinogen and other haemostasis parameters will serve as a surrogate measure of bleeding (and safety). In line with contemporary practice, investigators advise that patients have radial artery access whenever possible. Previous trials have used streptokinase (non-fibrin specific and immunogenic); this study will use the fibrin-specific non-immunogenic second generation thrombolytic, alteplase The only previous trial involved thrombolysis at the end of primary PCI (when microvascular thrombosis may already be established after reperfusion); the efficacy of thrombolysis may be greatest when thrombus is most abundant at the beginning of primary PCI; persistent residual fibrin strands adherent within the culprit territory will be selectively targeted by fibrinolytic therapy during primary PCI; thrombus which forms during the primary PCI procedure could be treated by the sustained 'deep tissue' thrombolytic effects of locally administered intra-coronary alteplase; in terms of ease-of-use and feasibility, there may be advantages to giving alteplase as a single dose.T-TIME is a Phase II evaluation of two reduced doses of alteplase, delivered locally, compared to placebo in STEMI patients receiving PCI in a double-blind, randomised, parallel group, placebo-controlled dose-ranging clinical trial. The investigators believe the strategy with intracoronary fibrinolysis complements other therapeutic approaches which are currently being tested. Should the trial demonstrate EFFICACY then a future trial might involve a factorial design with placebo, alteplase and any other intervention that might also be shown to be effective in the intervening time in order to test the comparative EFFICACY of each (alone or in combination) on surrogate and/or clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥ 18 years; females ≤ 18 years not of child bearing potential (defined as women who are post-menopausal or permanently sterilised (e.g. hysterectomy, tubal occlusion, bilateral salpingectomy)
* Acute myocardial infarction (symptoms onset ≤ 6 hours) with persistent ST-segment elevation or recent left bundle branch block
* Coronary artery occlusion (TIMI coronary flow grade 0 or 1) OR Impaired coronary flow (TIMI flow grade 2, slow but complete filling) in the presence of definite angiographic evidence of thrombus (TIMI grade 2+)
* Proximal-mid culprit lesion location in a major coronary artery (ie the right, left anterior descending, intermediate or circumflex coronary artery)
* Radial artery access

Exclusion Criteria:

* Shock (systolic blood pressure <90 mmHg with clinical signs of peripheral hypoperfusion despite adequate filling)
* Normal coronary flow grade (TIMI flow grade 3) at initial angiography
* Functional coronary collateral supply (Rentrop grade 2/3) to culprit artery
* Multivessel PCI intended before the day 2-7 MRI Scan
* Non-cardiac co-morbidity with expected survival <1 year
* Estimated body weight <60kg
* Contra-indication to contrast-enhanced MRI
* Pacemaker
* Implantable defibrillator
* estimated Glomerular Filtration Rate (eGFR) <30ml/min/1.73m²
* previous infarction in the culprit artery (known or suspected clinically, e.g. wall motion abnormality revealed by echocardiography)
* Significant bleeding problem either at present or within the past 6 months
* Patients with current concomitant oral anticoagulant therapy (INR > 1.3), including apixaban, dabigatran and rivaroxaban
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial, or spinal surgery)
* Known Haemorrhagic diathesis
* Severe uncontrolled hypertension >180/110 mmHg not controlled by medical therapy
* Major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with the current STEMI)
* Recent trauma to the head or cranium (<2 months)
* Prolonged cardiopulmonary resuscitation (>2 minutes) within past 2 weeks
* Acute pericarditis and/or subacute bacterial endocarditis e.g. valve mass or vegetation revealed by echocardiography
* Acute pancreatitis
* Severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis
* Arterial aneurysm and known arterial/venous malformation
* Neoplasm with increased bleeding risk
* Any known history of haemorrhagic stroke or stroke of unknown origin
* Known history of ischaemic stroke or transient ischaemic attack <6 months
* Dementia
* Hypersensitivity to gentamicin
* Women of child-bearing potential (i.e. pre-menopause) or breast feeding
* Previous randomisation to this study or participation in a study with an investigational drug or medical device within 90 days prior to randomisation
* Incapacity or inability to provide informed consent
* requirement for immunosuppressive drug therapy at any time during the past 3 months; whether administered orally, subcutaneously or intravenously. This would include corticosteroids (but not inhaled or topical), drugs used following transplantation (e.g. tacrolimus, cyclosporine), anti-metabolite therapies (e.g. mycophenolic acid (Myfortic), azathioprine, leflunomide (Arava)), and immunomodulators including biologics (e.g. adalimumab (HUMIRA), etanercept (Enbrel), aldesleukin), and DMARDS (cyclophosphamide. methotrexate, etc). Please note that this list is not exhaustive and a requirement for other immunosuppressive drugs not listed would also exclude the patient.
* active or prophylactic treatment with oral or parenteral antibiotic, antifungal or antiviral therapy to prevent or treat infection.
* any anti-cancer treatment (excluding surgery as this is covered above) at any time during the past 3 months including chemotherapy, radiotherapy and treatment with biologics such as Vascular Endothelial Growth Factor Receptor (VEGFR) inhibitors (e.g. bevacizumab, pazopanib). This list is not exhaustive and the sponsor or CI should be contacted for advice if required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
The amount of MVO (% of Left Ventricular (LV) mass) revealed by late (10 - 15 min) gadolinium contrast enhancement MRI 2 days post-MI. | 2-7 days
  Amount of MVO (% of LV mass) revealed by late gadolinium contrast-enhanced MRI 10-15 minutes after contrast administration on an MRI scan performed 2-7 days post-MI.

SECONDARY OUTCOMES:
Angiogram | 0-2 hours
  TIMI Coronary flow grade at the end of PCI; TIMI blush grade at the end of PCI; TIMI frame count at the end of PCI; TIMI thrombus grade at the end of PCI
ECG | 0-2 hours
  % ST segment resolution on the 12-lead ECG (pre- vs. 60 mins post-reperfusion with primary PCI)
Haematology | 24 hours
  Coagulation
MRI | 2-7 days
  Late MVO (presence/absence); Infarct size; Myocardial salvage index (infarct size/area-at-risk); LV end-diastolic volume (LVEDV); LV end-systolic volume (LVESV); LV ejection fraction (LVEF); Myocardial haemorrhage (presence/absence); Myocardial haemorrhage extent (% of LV)
Safety | 2-7 days
  Acute cerebral (stroke) and systemic (GI, peripheral) bleeding (if any) with alteplase; Coagulation (fibrinogen concentration);
MRI | 12 weeks
  Infarct size; Myocardial salvage index (final infarct size/initial area-at-risk); LV end-diastolic volume (LVEDV); LV end-systolic volume (LVESV); LV ejection fraction (LVEF);
ECG | 12 weeks
  ECG for final infarct size
Biochemistry | 12 weeks
  Troponin T; NT-pro BNP
Quality of Life | 12 weeks
  EQ5D-5L assessment (2-7 days, 12 weeks)

OTHER OUTCOMES:
Histopathology (sub-study) | 0 hours
  Fibrin histopathology in thrombus aspirate
Angiogram | 0-2 hours
  Intra-procedural changes in TIMI Coronary Flow Grade; Intra-procedural changes in TIMI blush grade; Intra-procedural changes in TIMI Frame Count; Intra-procedural changes in TIMI Thrombus Grade; Intra-procedural thrombotic events
Coronary Physiology (sub-study) | 0-2 hours
  IMR; CFR
Optical Coherence Tomography (sub-study) | 0-2 hours
  Thrombus area
Biochemistry | 24 hours
  Blood chemistry (standard of care blood tests)
Haematology | 24 hour
  Haemoglobin (standard of care blood tests)
Safety | 24 hours
  Haemoglobin (standard of care blood tests)
ECG | 12 weeks
  Surrogate ECG measures of infarct size - Anderson ST Acuteness score and Selvester QRS score; Acuteness of the ECG changes - Anderson Wilkins score;
MRI | 12 weeks
  First pass MVO extent (% of LV); Early MVO extent (% of LV) on 1 min post-gadolinium contrast enhanced MRI , adjusted for area-at-risk at baseline; LV remodelling index (minimum infarct wall thickness / maximum remote zone thickness mid-diastole); LV diastolic myocardial wall thickness to volume; LV sphericity index at end diastole (maximal longitudinal LV diameter (i.e. tip mitral valve to LV index) / maximal short-axis diameter); LV sphericity index at end-systole (maximal longitudinal LV diameter (i.e. tip mitral valve to LV apex) / maximal short-axis diameter); LV wall motion; Myocardial strain; Myocardial haemorrhage; Myocardial perfusion in the infarct zone; Myocardial perfusion in the remote zone; Infarct zone perfusion indexed to remote zone perfusion; Extracellular volume in the infarct zone; Extracellular volume in the remote zone; Extracellular in the infarct core; LV wall motion;
Quality of life | 2 years
  Blood chemistry (standard of care blood tests); EQ5D-5L (52 weeks)
Health outcomes | 3 years
  Death; MI; Heart Failure; Stroke/TIA; Acute bleeds

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, Prof, Principal Investigator — University of Glasgow
Locations (11):
- United Kingdom (11):
  - Edinburgh Royal Infirmary, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Leeds General Infirmary, Leeds
  - Glenfield Hospital, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Health Centre, St Bartholomew's Hospital, London
  - University Hospital of South Manchester NHS Foundation Trust, Manchester
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Heart and Lung Centre, New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Bulluck H, Carberry J, Carrick D, McCartney PJ, Maznyczka AM, Greenwood JP, Maredia N, Chowdhary S, Gershlick AH, Appleby C, Cotton JM, Wragg A, Curzen N, McEntegart M, Petrie MC, Eteiba H, Watkins S, Lindsay M, Mahrous A, Oldroyd KG, Berry C. A Noncontrast CMR Risk Score for Long-Term Risk Stratification in Reperfused ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Imaging. 2022 Mar;15(3):431-440. doi: 10.1016/j.jcmg.2021.08.006. Epub 2022 Jan 12. PMID 35272808
- [Derived] Maznyczka AM, McCartney PJ, Oldroyd KG, Lindsay M, McEntegart M, Eteiba H, Rocchiccioli JP, Good R, Shaukat A, Robertson K, Malkin CJ, Greenwood JP, Cotton JM, Hood S, Watkins S, Collison D, Gillespie L, Ford TJ, Weir RAP, McConnachie A, Berry C. Risk Stratification Guided by the Index of Microcirculatory Resistance and Left Ventricular End-Diastolic Pressure in Acute Myocardial Infarction. Circ Cardiovasc Interv. 2021 Feb;14(2):e009529. doi: 10.1161/CIRCINTERVENTIONS.120.009529. Epub 2021 Feb 16. PMID 33591821
- [Derived] Maznyczka AM, McCartney P, Duklas P, McEntegart M, Oldroyd KG, Greenwood JP, Muir D, Chowdhary S, Gershlick AH, Appleby C, Eteiba H, Cotton J, Wragg A, Curzen N, Tait RC, MacFarlane P, Welsh P, Sattar N, Petrie MC, Ford I, Fox KAA, McConnachie A, Berry C; T-TIME (Trial of low-dose adjunctive alTeplase during primary PCI) investigators. Effect of coronary flow on intracoronary alteplase: a prespecified analysis from a randomised trial. Heart. 2021 Jan 12:heartjnl-2020-317828. doi: 10.1136/heartjnl-2020-317828. Online ahead of print. PMID 33436493
- [Derived] Maznyczka AM, Oldroyd KG, Greenwood JP, McCartney PJ, Cotton J, Lindsay M, McEntegart M, Rocchiccioli JP, Good R, Robertson K, Eteiba H, Watkins S, Shaukat A, Petrie CJ, Murphy A, Petrie MC, Berry C. Comparative Significance of Invasive Measures of Microvascular Injury in Acute Myocardial Infarction. Circ Cardiovasc Interv. 2020 May;13(5):e008505. doi: 10.1161/CIRCINTERVENTIONS.119.008505. Epub 2020 May 15. PMID 32408817
- [Derived] McCartney PJ, Maznyczka AM, Eteiba H, McEntegart M, Oldroyd KG, Greenwood JP, Maredia N, Schmitt M, McCann GP, Fairbairn T, McAlindon E, Tait C, Welsh P, Sattar N, Orchard V, Corcoran D, Ford TJ, Radjenovic A, Ford I, McConnachie A, Berry C; T-TIME Investigators. Low-Dose Alteplase During Primary Percutaneous Coronary Intervention According to Ischemic Time. J Am Coll Cardiol. 2020 Mar 31;75(12):1406-1421. doi: 10.1016/j.jacc.2020.01.041. PMID 32216909
- [Derived] Maznyczka AM, Carrick D, Oldroyd KG, James-Rae G, McCartney P, Greenwood JP, Good R, McEntegart M, Eteiba H, Lindsay MM, Cotton JM, Petrie MC, Berry C. Thermodilution-derived temperature recovery time: a novel predictor of microvascular reperfusion and prognosis after myocardial infarction. EuroIntervention. 2021 Jun 25;17(3):220-228. doi: 10.4244/EIJ-D-19-00904. PMID 32122822
- [Derived] Maznyczka AM, McCartney PJ, Oldroyd KG, Lindsay M, McEntegart M, Eteiba H, Rocchiccioli P, Good R, Shaukat A, Robertson K, Kodoth V, Greenwood JP, Cotton JM, Hood S, Watkins S, Macfarlane PW, Kennedy J, Tait RC, Welsh P, Sattar N, Collison D, Gillespie L, McConnachie A, Berry C. Effects of Intracoronary Alteplase on Microvascular Function in Acute Myocardial Infarction. J Am Heart Assoc. 2020 Feb 4;9(3):e014066. doi: 10.1161/JAHA.119.014066. Epub 2020 Jan 28. PMID 31986989
- [Derived] McCartney PJ, Eteiba H, Maznyczka AM, McEntegart M, Greenwood JP, Muir DF, Chowdhary S, Gershlick AH, Appleby C, Cotton JM, Wragg A, Curzen N, Oldroyd KG, Lindsay M, Rocchiccioli JP, Shaukat A, Good R, Watkins S, Robertson K, Malkin C, Martin L, Gillespie L, Ford TJ, Petrie MC, Macfarlane PW, Tait RC, Welsh P, Sattar N, Weir RA, Fox KA, Ford I, McConnachie A, Berry C; T-TIME Group. Effect of Low-Dose Intracoronary Alteplase During Primary Percutaneous Coronary Intervention on Microvascular Obstruction in Patients With Acute Myocardial Infarction: A Randomized Clinical Trial. JAMA. 2019 Jan 1;321(1):56-68. doi: 10.1001/jama.2018.19802. PMID 30620371